CLINICAL TRIAL: NCT02173470
Title: Ultra Low-dose Chest CT With Iterative Reconstructions as an Alternative to Conventional Chest X-ray Prior to Heart Surgery
Brief Title: Chest CT With Iterative Reconstruction as an Alternative to Conventional Chest X-ray Prior to Heart Surgery
Acronym: CRICKET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Expected futility in reaching the primary endpoint
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Annemarie den Harder, MD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL47293.041.13; 837001403 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2014-06-17; First posted 2014-06-25 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Cardiac Defects; Disorder; Heart, Functional, Postoperative, Cardiac Surgery; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Routine clinical care (which includes a conventional chest X-ray).
- CT scan (Experimental): Routine clinical care, which includes a chest x-ray, with an additional ultra low-dose non contrast enhanced chest CT with IR (performed preoperatively).
  Interventions: Other: CT scan

INTERVENTIONS:
Other: CT scan — The intervention group receives both standard care (chest x-ray) and an ultra low dose CT thorax without contrast.
  Other Names: computed tomography
  Arms: CT scan

SUMMARY:
To assess if information about aortic calcification obtained from routine preoperative ultra low-dose chest CT lowers the postoperative stroke rate in patients undergoing heart surgery by optimizing surgical strategy compared to the normal work-up with a conventional chest X-ray.

DETAILED DESCRIPTION:
During heart surgery the aorta is clamped to initiate cardiopulmonary bypass. This may crush aortic calcifications causing them to embolize to the brain causing a stroke which is a devastating complication for the patient. A chest X-ray is routinely performed prior to heart surgery. It provides no information about aortic calcification. Imaging by a chest computed tomography (CT) scan provides detailed information on aortic calcification but has higher radiation exposure and thus is not used routinely. Recently iterative reconstruction (IR) techniques have become available that allow chest CT to be performed at markedly reduced dose with retained image quality. Routine use of low dose chest CT with IR prior to heart surgery may identify patients with a severely calcified aorta in which the surgery may subsequently adapted to minimize or avoid aortic manipulation which may reduce stroke rate.

In this multicenter randomized controlled clinical trial the effect of preoperative chest CT on postoperative stroke is investigated. In total 1724 patients will be included of whom 862 patients will receive an additional CT to standard care and 862 patients will receive routine care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Scheduled to undergo heart surgery
* Provide written informed consent

Exclusion Criteria:

* Patient not meeting inclusion criteria
* Pregnant women
* Scheduled to undergo transcatheter aortic valve insertion procedure (since these patients receive a standard preoperative CT)
* Chest or cardiac CT in the past three months
* Emergency surgery
* Concomitant or previous participation in a study that prohibits the patient from participating in a study that exposed the patient to radiation
* Unwillingness to be informed about unrequested findings on the CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 866 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Postoperative stroke | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  Percentage of patients suffering from in-hospital postoperative stroke (central neurological defect that either recovers spontaneously or is permanent) after heart surgery.

SECONDARY OUTCOMES:
Altered surgical approach | The surgery will take place the day after hospital administration.
  Percentage of patients in which the surgical approach is altered based on information derived from the preoperative chest CT.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo PJ Budde, MD, PhD, Principal Investigator — Erasmus MC Rotterdam
Locations (3):
- Heart and Vascular Center Semmelweis University, Budapest, Hungary
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- Available data/document: Study Protocol — http://www.ncbi.nlm.nih.gov/pubmed/26857421 — Ultra low-dose chest ct with iterative reconstructions as an alternative to conventional chest x-ray prior to heart surgery (CRICKET study): Rationale and design of a multicenter randomized trial.